CLINICAL TRIAL: NCT06087588
Title: The Impact of the Pericapsular Nerve Group Block (PENG) Chemical Neurolysis on the Quality of Life of Patients with Advanced Hip Osteoarthritis. a Randomized, Prospective Double-blinded Clinical Trial.
Brief Title: Pericapsular Nerve Group Block Chemical Neurolysis in Advanced Hip Osteoarthritis
Acronym: PENG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5/2023
Record Dates: First submitted 2023-07-05; First posted 2023-10-18 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip | interventions — Sodium Chloride; Ethanol; Nerve Block

STUDY DESIGN:
Intervention Model Description: Group 1 - PENG sham block Group 2 - PENG neurolysis 95% ethanol
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sham PENG block (Active Comparator): PENG block - 20ml 0,9% normal saline
  Interventions: Drug: 0.9%sodium chloride
- PENG neurolysis (Active Comparator): PENG neurolysis with 5ml 95% ethanol
  Interventions: Drug: 95% ethanol

INTERVENTIONS:
Drug: 0.9%sodium chloride — PENG sham block with 20ml 0,9% normal saline
  Other Names: Sham block
  Arms: sham PENG block
Drug: 95% ethanol — PENG neurolysis with 2.5ml of 95% ethanol
  Other Names: neurolysis
  Arms: PENG neurolysis

SUMMARY:
PENG neurolysis in advanced osteoarthritis of the hip joint.

DETAILED DESCRIPTION:
The study aims to assess the safety and effectiveness of regional pain treatment methods and their impact on the quality of life of patients with advanced osteoarthritis of the hip joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Pain Treatment Clinic of the Transfiguration of Jesus Clinical Hospital of the Medical University of Poznań will be qualified for the study
* patients with coxarthrosis or gonarthrosis who failed to achieve satisfactory pain control (NRS>3) despite the use of NSAIDs, Paracetamol, and co-analgetics
* Age of patients: from 18 to 110 years of age.
* Caucasian patients can give informed, complete, written consent.

Exclusion Criteria:

* suspected or diagnosed opioid dependence syndrome
* active cancer
* dementia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
NRS score | 7 days after procedure
  The NRS (Numeric Pain Rating Scale) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
NRS score | 30 days after procedure
  The NRS (Numeric Pain Rating Scale) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
NRS score | 3 months after procedure
  The NRS (Numeric Pain Rating Scale) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
NRS score | 6 months after procedure
  The NRS (Numeric Pain Rating Scale) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.

SECONDARY OUTCOMES:
Health Questionnaire (EQ-5D-5L) | 7 days after procedure
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
Health Questionnaire (EQ-5D-5L) | 30 days after procedure
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
Health Questionnaire (EQ-5D-5L) | 3 months after procedure
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
Health Questionnaire (EQ-5D-5L) | 6 months after procedure
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
neurological deficits | 7 days after procedure
  yes/no
neurological deficits | 30 days after procedure
  yes/no
neurological deficits | 3 months after procedure
  yes/no
neurological deficits | 6 months after procedure
  yes/no
total opioid consumption | 7 days after procedure
  milligrams of oral morphine per day
total opioid consumption | 30 days after procedure
  milligrams of oral morphine per day
total opioid consumption | 3 months after procedure
  milligrams of oral morphine per day
total opioid consumption | 6 months after procedure
  milligrams of oral morphine per day

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Wieczorowska-Tobis, Prof.dr hab, Study Director — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reysner M, Reysner T, Kowalski G, Mularski A, Daroszewski P, Wieczorowska-Tobis K. Chemical ablation of pericapsular nerve group with 95% ethanol for pain relief and quality of life in patients with hip osteoarthritis: a prospective, double-blinded, randomised, controlled trial. Br J Anaesth. 2025 Aug;135(2):382-389. doi: 10.1016/j.bja.2025.04.045. Epub 2025 Jun 6. PMID 40480912